CLINICAL TRIAL: NCT04497779
Title: Evaluation of Coronavirus Disease 19 (COVID-19) Convalescent Plasma
Brief Title: Analysis of Coronavirus Disease 19 (COVID-19) Convalescent Plasma
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Other Study IDs: 20204; NCI-2020-04000 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20204 (Other: City of Hope Medical Center); P30CA033572 (NIH); TGen (Other: Translational Genomics Research Institute (TGen))
Record Dates: First submitted 2020-06-29; First posted 2020-08-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Asymptomatic COVID-19 Infection Laboratory-Confirmed; Symptomatic COVID-19 Infection Laboratory-Confirmed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab, blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Screening (biospecimen collection, medical record review, CCP): PROSPECTIVE CCP DONORS: Participants undergo collection of blood and/or nasopharyngeal swabs at the time of screening. Participants' medical records are reviewed.
  CONVALESCENT BLOOD DONORS WHO CHOOSE NOT TO DONATE CCP: Participants undergo collection of blood sample at the time of screening. Participants' medical records are reviewed.
  CCP RECIPIENTS: Patients undergo collection of blood samples at baseline, 12-24 hours after each CCP infusion, and 7 days after last CCP infusion. Patients' medical records are reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Diagnostic Laboratory Biomarker Analysis; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and/or nasopharyngeal swabs
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Other: Electronic Health Record Review — Donors and recipients have their medical records reviewed.
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
Plasma from patients who have recovered from coronavirus disease 2019 (COVID-19) is referred to as COVID-19 convalescent plasma (CCP), and may contain antibodies against SARS-CoV-2, the virus responsible for COVID-19. CCP infusion is being evaluated as a therapeutic or prophylactic approach in COVID-19 patients. The goal of this study is to help develop a bank of convalescent plasma in California, especially in medically underserved communities particularly affected by the disease. In parallel, CCP administered to COVID-19 patients will be collected and analyzed to determine whether the antibody profile correlates with clinical outcome. The purpose of this non-therapeutic study is to learn more about the CCP antibody profile and the effect it may have in treating COVID-19 infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish a testing service for screening prospective donors of coronavirus disease 2019 (COVID-19) convalescent plasma (CCP).

II. Characterize the titer and neutralizing properties of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) antibodies in CCP.

III. Correlate the SARS-CoV-2 antibody characteristics in CCP with the outcome in severely ill COVID-19 patients treated with CCP.

EXPLORATORY OBJECTIVES:

I. Facilitate the recruitment of CCP donors in medically underserved areas.

II. Develop high-throughput methods for detection/characterization of SARS-CoV-2 neutralizing and non-neutralizing antibodies.

III. Develop a bank of convalescent plasma that would be available for future studies relating to the content of CCP.

IV. Study the impact of antibody levels, donor characteristics and patient characteristics on outcome in COVID-19 patients treated with CCP.

V. Procure blood samples from COVID-19 convalescent volunteers for future COVID-19-related studies.

OUTLINE:

PROSPECTIVE CCP DONORS: Participants undergo collection of blood and/or nasopharyngeal swabs at the time of screening. Participants' medical records are reviewed.

CONVALESCENT BLOOD DONORS WHO CHOOSE NOT TO DONATE CCP: Participants undergo collection of blood sample at the time of screening. Participants' medical records are reviewed.

CCP RECIPIENTS: Patients undergo collection collection of blood samples at baseline, between CCP unit infusions, 24 hours after last CCP infusion, and between 14-28 after last CCP infusion. Patients' medical records are reviewed.

ELIGIBILITY:
For COVID-19 convalescent individuals:

* Age: ≥ 18 years
* Evidence of COVID-19 documented by a laboratory test either by: a diagnostic test (e.g., a NP swab) at the time of illness OR a positive serological test for SARS-CoV-2 antibodies after recovery, if prior diagnostic testing was not performed at the time COVID-19 was suspected.

Note: If volunteers can't provide evidence of COVID-19, but are otherwise eligible, then we will test them for SARS-CoV-2 antibodies to confirm eligibility.

* Be willing to complete a pre-screening questionnaire
* Be willing to donate blood samples
* Permit medical record review
* For prospective CCP donors only: weigh more than 110 pounds and be in general good health

For (COVID-19 convalescent plasma (CCP) recipients:

* Be enrolled in a clinical trial involving the infusion of CCP for the treatment of COVID-19.
* Be willing to provide blood samples
* Permit medical record review

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosis of laboratory-confirmed COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
Convalescent plasma (CCP) units infused in coronavirus disease-2019 (COVID-19) patients | Up to 12 months after enrollment
  Will be assayed for severe acute respiratory syndrome (SARS-CoV-2) immunoassay, coronavirus (CoV) PepSeq assay, and SARS-CoV-2 lenti-based neutralizing antibody titer.
All-cause mortality | At day 28 post-CCP infusion
  Will naturally be compared to reported data from the other studies. Analysis will focus on demonstrating that the antibody content of donor plasma increases the odds of surviving past day 28. Will also develop a nomogram for the probability of success (alive at day 28), accounting for patient, donor material and donor antibody characteristics measurable covariates.
Donor antibody levels | Up to 28 days post-CCP infusion
  Will be examined to see how this relates to the duration of hospitalization.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 28 days post-CCP infusion
  Will be assessed on a 7-point ordinal scale, as recommended by the WHO patient outcome R&D Blueprint Group.
CCP recipient outcomes | Up to 28 days post-CCP infusion
  Will be assessed on a 7-point ordinal scale. The scale is as follows:
  1. Death;
  2. Hospitalized, on invasive mechanical ventilation or ECMO;
  3. Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  4. Hospitalized, requiring low flow supplemental oxygen;
  5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise);
  6. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care (other than per protocol RDV administration);
  7. Not hospitalized

OTHER OUTCOMES:
Duration of hospitalization (days) | Up to 28 days post-CCP infusion
  Patient can stay at the hospital for up to 28 days post-CCP infusion
Time to clinical improvement (days) | Up to 28 days post-CCP infusion
  Will be assessed on a 7-point ordinal scale.

CONTACTS AND LOCATIONS:
Overall Officials: John Zaia, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States